CLINICAL TRIAL: NCT04094506
Title: A Phase 1, Open-label Study of ASP1948, Targeting an Immune Modulatory Receptor, in Japanese Patients With Advanced Solid Tumors
Brief Title: Study of ASP1948, Targeting an Immune Modulatory Receptor, in Japanese Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1948-CL-0102
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Locally Advanced (Unresectable) or Metastatic Solid Tumor Malignancies
Keywords: safety; ASP1948; pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- ASP1948 1200 mg (Experimental): Participants received 1200 mg ASP1948 intravenously, on day 1 of cycle 1 and 2 followed by once every 2 weeks (Q2W) until discontinuation criteria or up to 2 years. Each cycle duration was 14 days.
  Interventions: Drug: ASP1948
- ASP1948 2000 mg (Experimental): Participants received 2000 mg ASP1948 intravenously, on day 1 of cycle 1 and 2 followed by once Q2W until discontinuation criteria or up to 2 years. Each cycle duration was 14 days.
  Interventions: Drug: ASP1948
- ASP1948 3000 mg (Experimental): Participants received 3000 mg ASP1948 intravenously, on day 1 of cycle 1 followed by once every 3 weeks until discontinuation criteria or up to 2 years. Each cycle duration was 21 days.
  Interventions: Drug: ASP1948

INTERVENTIONS:
Drug: ASP1948 — Intravenous

SUMMARY:
The primary purpose of this study is to evaluate the tolerability, safety and pharmacokinetic profile of ASP1948 in Japanese patients with locally advanced (unresectable) or metastatic solid tumors.

This study will also evaluate the antitumor effect of ASP1948.

DETAILED DESCRIPTION:
This study consists of 3 dose levels (1200 milligrams [mg], 2000 mg and 3000 mg) and enrollment of subjects into dose level 1200 mg will take place first. Dose level 2000 mg would only be opened if dose level 1200 mg is deemed tolerable. Dose level 3000 mg would only be opened if dose level 2000 mg is deemed tolerable.

ELIGIBILITY:
Inclusion Criteria:

* Subject has locally advanced (unresectable) or metastatic solid tumor malignancy (no limit to the number of prior treatment regimens) that is confirmed by available pathology records or current biopsy (if needed) and has received all standard therapies (unless the therapy is contraindicated or intolerable) felt to provide clinical benefit for his/her specific tumor type.
* Subject has an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Subject's last dose of prior antineoplastic therapy, including any immunotherapy, was at least 21 days prior to initiation of investigational product (IP) administration. A subject with epidermal growth factor receptor (EGFR) or anaplastic lymphoma kinase (ALK) mutation-positive non-small cell lung cancer (NSCLC) is allowed to remain on EGFR tyrosine kinase inhibitor (TKI) or ALK inhibitor therapy until 4 days prior to initiation of IP administration.
* Subject has completed any radiotherapy (including stereotactic radiosurgery) at least 14 days prior to initiation of IP administration.
* Subject with metastatic castration resistant prostate cancer (mCRPC) (positive bone scan and/or soft tissue disease documented by computed tomography [CT]/magnetic resonance imaging [MRI]) meets both of the following:

  * Subject has serum testosterone ≤ 50 ng/dL at Screening.
  * Subject has had an orchiectomy or plans to continue androgen deprivation therapy (ADT) for the duration of study treatment.
* Subject has adequate organ function as indicated by laboratory values within 7 days prior to initiation of IP administration. (If a subject has received a recent blood transfusion, the laboratory tests must be obtained ≥ 28 days after any blood transfusion.) Note: Growth factors, colony stimulating factors are not permitted in the screening period.
* Female subject is not pregnant and at least 1 of the following conditions apply:

  * Not a woman of childbearing potential (WOCBP)
  * WOCBP who agrees to follow the contraceptive guidance from the time of informed consent throughout the treatment period and for at least 6 months after the final study treatment administration.
* Female subject must agree not to breastfeed starting at Screening and throughout the study period, and for 6 months after the final study treatment administration.
* Female subject must not donate ova starting at first dose of IP and throughout the study period, and for 6 months after the final study treatment administration.
* Male subject with female partner(s) of childbearing potential (including breastfeeding partner) must agree to use contraception throughout the treatment period and for at least 6 months after the final study treatment administration.
* Male subject must not donate sperm during the treatment period and for 6 months after the final study treatment administration.
* Male subject with a pregnant partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy throughout the study period and for 6 months after the final study treatment administration.
* Subject agrees not to participate in another interventional study while receiving study treatment in the present study (subjects who are currently in the follow-up period of an interventional clinical study are allowed).

Exclusion Criteria:

* Subject weighs < 45 kg at Screening.
* Subject has received investigational therapy within 21 days prior to start of IP. (A subject with EGFR activating mutations or a subject with an ALK mutation is allowed to remain on an investigational EGFR TKI or ALK inhibitor until 4 days prior to initiation of IP administration.)
* Subject requires or has received systemic steroid therapy or any other immunosuppressive therapy within 14 days prior to IP administration. Subjects using a physiologic replacement dose of hydrocortisone or its equivalent (defined as up to 30 mg per day of hydrocortisone, 2 mg per day of dexamethasone or up to 10 mg per day of rednisone) are allowed. Note: corticosteroids for prophylaxis (e.g., contrast dye allergy) or for brief treatment of conditions not related to study treatment (e.g., delayed-type hypersensitivity reaction caused by a contact allergen) is also allowed.
* Subject has symptomatic central nervous system (CNS) metastases or subject has evidence of unstable CNS metastases even if asymptomatic (e.g., progression on scans). Subjects with previously treated CNS metastases are eligible, if they are clinically stable and have no evidence of CNS progression by imaging for at least 28 days prior to start of study treatment and are not requiring immunosuppressive doses of systemic steroids (> 30 mg per day of hydrocortisone, > 2 mg per day of dexamethasone or > 10 mg per day of prednisone or equivalent) for longer than 14 days.
* Subject has leptomeningeal disease as a manifestation of the current malignancy.
* Subject has an active autoimmune disease. Subjects with type 1 diabetes mellitus, stable endocrinopathies maintained on appropriate replacement therapy and skin disorders (e.g., vitiligo, psoriasis or alopecia) not requiring systemic treatment are allowed.
* Subject was discontinued from prior immunomodulatory therapy due to a Grade ≥ 3 toxicity that was mechanistically related (e.g., immune-related) to the agent.
* Subject has known history of serious hypersensitivity reaction to a known ingredient of ASP1948 or severe hypersensitivity reaction to treatment with another monoclonal antibody.
* Subject is positive for Hepatitis B virus (HBV) antibodies and surface antigen (including acute HBV or chronic HBV) or Hepatitis C virus ([HCV] ribonucleic acid [RNA]). Hepatitis C RNA testing is not required in subjects with negative Hepatitis C antibody testing. HBV antibodies are not required in subjects with negative Hepatitis B surface antigen (HBsAg).
* Subject has received a live vaccine against infectious diseases within 28 days prior to initiation of study treatment.
* Subject has a history of drug-induced pneumonitis (interstitial lung disease) or currently has pneumonitis.
* Subject has an active infection requiring systemic therapy (e.g., intravenous antibiotics) within 14 days prior to IP treatment.
* Subject is expected to require another form of antineoplastic therapy while on study treatment.
* Subject has an uncontrolled intercurrent illness including, but not limited to cardiac arrhythmia or psychiatric illness/social situations that would limit compliance with study requirements.
* Subject's AEs (excluding alopecia) from prior therapy have not improved to Grade 1 or baseline within 14 days prior to start of study treatment.
* Subject has significant cardiovascular disease including:

  * Subject has inadequately controlled hypertension (defined as systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg on antihypertensive medications).
  * Subject has a history of myocardial infarction or unstable angina within 6 months prior to Cycle 1 Day 1.
  * Subject has New York Heart Association Class II or greater chronic heart failure.
  * History of cerebrovascular accident (CVA) or transient ischemic attack (TIA) within 6 months prior to study treatment.
  * Subject has significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to study treatment.
* Subject has a history of hemoptysis (bright red blood of 2 mL or more per episode) within 12 weeks prior to study treatment.
* Subject has evidence of a bleeding diathesis or significant coagulopathy.
* Subject has inadequate recovery from prior surgical procedure or has had a major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to study treatment, or anticipates the need for a major surgical procedure during the course of the study or minor surgery within 7 days of starting study treatment.
* Subject has initiated new treatment with medications that affect the coagulation cascade with international normalized ratio (INR) ≥ 2 such as vitamin K antagonists, heparins and direct thrombin inhibitors or the use of factor Xa inhibitors within 28 days prior to the start of study treatment. Note: If the subject started receiving such medications more than 28 days prior to the start of study treatment and needs to continue, this is allowed. However, new anticoagulation may not be initiated within 28 days prior to the start of study treatment.
* Subject has any condition that makes the subject unsuitable for study participation.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2022-02-02 (Actual); Study Completion 2022-02-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with Dose Limiting Toxicity (DLT) for Dose level 1200 mg and 2000 mg | Up to 28 days
  DLT is graded using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 4.03. The DLT observation period may be increased if deemed appropriate by Dose Escalation and Safety Committee.
Number of participants with DLT for Dose level 3000 mg | Up to 21 days
  DLT is graded using NCI-CTCAE Version 4.03. The DLT observation period may be increased if deemed appropriate by Dose Escalation and Safety Committee.
Number of participants with Adverse Events (AEs) | Up to 30 days after the final IP administration or initiation of a new anticancer treatment, whichever comes first (a maximum of 108 weeks)
  An AE is any untoward medical occurrence in a subject administered an investigational product (IP) and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of IP whether or not considered related to the IP.
Number of participants with immune-related AEs (irAEs) | Up to 30 days after the final IP administration or initiation of a new anticancer treatment, whichever comes first (a maximum of 108 weeks)
  Number of participants with potentially clinically significant irAEs. irAEs observed with currently approved checkpoint inhibitors (CPIs) include rash, oral mucositis, dry mouth, colitis/diarrhea, hepatitis, pneumonitis and endocrinopathies (hypophysitis, hypothyroidism, hyperthyroidism, adrenal insufficiency and Type 1 diabetes mellitus).
Number of participants with infusion-related reactions (IRRs) | Up to 30 days after the final IP administration or initiation of a new anticancer treatment, whichever comes first (a maximum of 108 weeks)
  Number of participants with potentially clinically significant IRRs. The majority of IRRs to monoclonal antibodies represent "standard" infusion reactions, and the most common manifestations of these standard infusion reactions include: fever and/or shaking/chills; flushing and/or itching; changes in heart rate and blood pressure; shortness of breath or chest discomfort; pain in back or abdomen; nausea, vomiting and/or diarrhea and skin rash (various types). Fever and muscle pain suggest that the reaction is a standard infusion reaction.
Number of participants with serious AEs (SAEs) | Up to 90 days after the final IP administration or initiation of a new anticancer treatment, whichever comes first (a maximum of 116 weeks)
  Adverse event (AE) is considered "serious" if the investigator or sponsor view any of the following outcomes: Death, life-threatening, persistent or significant disability/incapacity, congenital anomaly or birth defect, hospitalization, or medically important event.
Number of participants with complete blood count (CBC) value abnormalities and/or AEs | Up to 30 days after the final IP administration or initiation of a new anticancer treatment, whichever comes first (a maximum of 108 weeks)
  Number of participants with potentially clinically significant CBC values.
Number of participants with serum chemistry value abnormalities and/or AEs | Up to 30 days after the final IP administration or initiation of a new anticancer treatment, whichever comes first (a maximum of 108 weeks)
  Number of participants with potentially clinically significant serum chemistry values.
Number of participants with urinalysis value abnormalities and/or AEs | Up to end of treatment period (a maximum of 104 weeks)
  Number of participants with potentially clinically significant urinalysis values.
Number of participants with prothrombin time/international normalized ratio (PT/INR) value abnormalities and/or AEs | Up to 30 days after the final IP administration or initiation of a new anticancer treatment, whichever comes first (a maximum of 108 weeks)
  Number of participants with potentially clinically significant PT/INR values.
Number of participants with activated partial thromboplastin time (aPTT) value abnormalities and/or AEs | Up to 30 days after the final IP administration or initiation of a new anticancer treatment, whichever comes first (a maximum of 108 weeks)
  Number of participants with potentially clinically significant aPTT values.
Number of participants with thyroid stimulating hormone (TSH) value abnormalities and/or AEs | Up to 30 days after the final IP administration or initiation of a new anticancer treatment, whichever comes first (a maximum of 108 weeks)
  Number of participants with potentially clinically significant TSH values.
Number of participants with free thyroxine (free T4) value abnormalities and/or AEs | Up to 30 days after the final IP administration or initiation of a new anticancer treatment, whichever comes first (a maximum of 108 weeks)
  Number of participants with potentially clinically significant free T4 values.
Number of participants with electrocardiogram (ECG) abnormalities and/or AEs | Up to end of treatment period (a maximum of 104 weeks)
  Number of participants with potentially clinically significant ECG values.
Number of participants with vital sign abnormalities and/or AEs | Up to 90 days after the final IP administration or initiation of a new anticancer treatment, whichever comes first (a maximum of 116 weeks)
  Number of participants with potentially clinically significant vital sign values.
Number of participants with physical exams abnormalities and/or AEs | Up to end of treatment period (a maximum of 104 weeks)
  Number of participants with potentially clinically significant physical exams values.
Eastern Cooperative Oncology Group (ECOG) performance status score | Up to 30 days after the final IP administration or initiation of a new anticancer treatment, whichever comes first (a maximum of 108 weeks)
  The ECOG scale will be used to assess performance status. Grades range from 0 (fully active) to 4 (completely disabled). Negative change scores indicate an improvement. Positive scores indicate a decline in performance.
Pharmacokinetics (PK) of ASP1948 in serum: Area under the concentration-time curve (AUC) from the time of dosing to the last measurable concentration (AUClast) | Up to 90 days after the final IP administration or initiation of a new anticancer treatment, whichever comes first (a maximum of 116 weeks)
  AUClast will be recorded from the PK serum samples collected.
PK of ASP1948 in serum: AUC from the time of dosing extrapolated to time infinity (AUCinf) | Up to 90 days after the final IP administration or initiation of a new anticancer treatment, whichever comes first (a maximum of 116 weeks)
  AUCinf will be recorded from the PK serum samples collected.
PK of ASP1948 in serum: Percentage of AUCinf due to extrapolation from the last measurable concentration to time infinity (AUCinf(%extrap)) | Up to 90 days after the final IP administration or initiation of a new anticancer treatment, whichever comes first (a maximum of 116 weeks)
  AUCinf(%extrap) will be recorded from the PK serum samples collected.
PK of ASP1948 in serum: AUC from the time of dosing to the start of next dosing interval (AUCtau) | Up to 90 days after the final IP administration or initiation of a new anticancer treatment, whichever comes first (a maximum of 116 weeks)
  AUCtau will be recorded from the PK serum samples collected.
PK of ASP1948 in serum: maximum concentration (Cmax) | Up to 90 days after the final IP administration or initiation of a new anticancer treatment, whichever comes first (a maximum of 116 weeks)
  Cmax will be recorded from the PK serum samples collected.
PK of ASP1948 in serum: concentration immediately prior to dosing at multiple dosing (Ctrough) | Up to 90 days after the final IP administration or initiation of a new anticancer treatment, whichever comes first (a maximum of 116 weeks)
  Ctrough will be recorded from the PK serum samples collected.
PK of ASP1948 in serum: dosing time of maximum concentration (tmax) | Up to 90 days after the final IP administration or initiation of a new anticancer treatment, whichever comes first (a maximum of 116 weeks)
  tmax will be recorded from the PK serum samples collected.
PK of ASP1948 in serum:dosing: terminal elimination half-life (t1/2) | Up to 90 days after the final IP administration or initiation of a new anticancer treatment, whichever comes first (a maximum of 116 weeks)
  t1/2 will be recorded from the PK serum samples collected.
PK of ASP1948 in serum: time of last measurable concentration (tlast) | Up to 90 days after the final IP administration or initiation of a new anticancer treatment, whichever comes first (a maximum of 116 weeks)
  tlast will be recorded from the PK serum samples collected.
PK of ASP1948 in serum: total clearance after intravenous dosing (CL) | Up to 90 days after the final IP administration or initiation of a new anticancer treatment, whichever comes first (a maximum of 116 weeks)
  CL will be recorded from the PK serum samples collected.
PK of ASP1948 in serum: volume of distribution after intravenous dosing (V) | Up to 90 days after the final IP administration or initiation of a new anticancer treatment, whichever comes first (a maximum of 116 weeks)
  V will be recorded from the PK serum samples collected.

SECONDARY OUTCOMES:
Percent change in tumor size from baseline | Up to end of treatment period (a maximum of 104 weeks)
  Tumor size is defined as the sum of the diameters of all target lesions per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. The percent change from baseline in tumor size will be calculated for subjects with target lesions at baseline. The best percent change in tumor size is the maximum percent reduction from baseline, or if the subject has no reduction in size, the minimum percent increase from baseline.
Number of participants with best overall response (BOR)per RECIST 1.1 and 'immune' Response Evaluation Criteria in Solid Tumors (iRECIST) | Up to end of treatment period (a maximum of 104 weeks)
  BOR is defined as the best response recorded from the start of the study treatment until the end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma Inc
Locations (1):
- Site JP810001, Chuo-ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website — https://www.clinicaltrials.astellas.com/study/1948-CL-0102/
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=14522&tenant=MT_AST_9011